CLINICAL TRIAL: NCT04350892
Title: Changes in Cerebrospinal Fluid Biomarkers After Bariatric Surgery
Brief Title: Cerebrospinal Fluid Biomarkers in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sharon Wardlaw, Dr. Robert C. and Veronica Atkins Professor of Obesity Research, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS8430; 1R01DK124465 (NIH)
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Obesity; Bariatric Surgery; Gastric Bypass; Sleeve Gastrectomy; Weight Loss; Low Calorie Diet
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Roux-en-Y Gastric Bypass Surgery (Active Comparator)
  Interventions: Procedure: Roux-en-Y Gastric Bypass (RYGB)
- Sleeve Gastrectomy Surgery (Active Comparator)
  Interventions: Procedure: Sleeve Gastrectomy (SG)
- Very Low Calorie Diet (Active Comparator)
  Interventions: Behavioral: Very Low Calorie Diet (VLCD)

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass (RYGB) — This surgery is often called gastric bypass. It is a weight-loss surgery that involves creating a small stomach pouch and bypassing part of the small intestine.
  If you decide with your doctor to have gastric bypass, you can be enrolled on this arm of the study. A surgery date should be pending before the investigators screen you for the study. The study does not cover the cost of the Roux-en-Y gastric bypass.
  Arms: Roux-en-Y Gastric Bypass Surgery
Procedure: Sleeve Gastrectomy (SG) — Sleeve gastrectomy, is a weight-loss surgery that involves removing about 80% of the stomach.
  If you decide with your doctor to have sleeve gastrectomy, you can be enrolled on this arm of the study. A surgery date should be pending before the investigators screen you for the study. The study does not cover the cost of the sleeve gastrectomy.
  Arms: Sleeve Gastrectomy Surgery
Behavioral: Very Low Calorie Diet (VLCD) — Weight loss with calorie restricted liquid diet. Participants will be placed on a 800 kcal/day diet for meal replacement (Optifast) provided by the investigator for 12 weeks. Participants will be monitored weekly by the study dietician and medical staff.
  Arms: Very Low Calorie Diet

SUMMARY:
The goal of this project is to understand why bariatric surgery is such an effective treatment for obesity with a focus on brain mechanisms. Cerebrospinal fluid (CSF) neuropeptide, hormone and protein levels will be measured as a surrogate for changes in brain activity in participants before and after bariatric surgery as compared with participants before and after diet-induced weight loss. The investigators are studying neuropeptides and hormones that are know to be involved with the regulation of appetite and body weight to determine if some of the changes that are expected to occur after diet-induced weight loss do not occur after bariatric surgery. In addition, proteomic analysis will be used to uncover new protein biomarkers that are unique to surgical weight loss. The results of these studies will help explain why bariatric surgery is so effective in achieving long-term weight loss. Understanding how the central nervous system responds to bariatric surgery could help the development of alternative nonsurgical therapies for obesity and its metabolic complications.

DETAILED DESCRIPTION:
Peripheral metabolic signals communicate levels of energy stores to the brain and elicit a host of neuronal responses that maintain energy balance; such regulatory mechanisms make it difficult to maintain diet-induced weight loss. The goal is to understand how these central regulatory mechanisms are circumvented following surgical alterations in the gut in subjects after Roux-en-Y gastric bypass (RYGB) and vertical sleeve gastrectomy (SG) compared to carefully matched diet- induced weight loss controls who achieve weight loss on a low calorie liquid diet. Surgery participants will be patients who have already chosen to have a bariatric surgery procedure with their doctor. Diet participants will be provided with the low calorie liquid diet for approximately 3 months and will be monitored weekly throughout the study.

Surgery participants will be studied at 3 time-points:

1. Before the intervention
2. After surgery at 10-15% weight loss
3. At 12 months after surgery

Low calorie diet participants will be studied at 2 time-points:

1. Before intervention
2. At 10-15% weight loss (approximately 12 weeks on the diet)

At each time-point subjects will have a lumbar puncture (spinal tap) for cerebrospinal fluid (CSF) sampling and blood will be collected in the fasting state and in response to a liquid meal challenge. Body weight, waist and hip circumference will be measured.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* BMI 35-55

Exclusion Criteria:

* No clinically significant medical conditions
* No use of tobacco
* No alcohol or drug abuse
* No recent weight change (+/-5%) within prior 6 months
* No medications that may affect body weight or blood glucose
* No diabetes medications, beta-blockers, opiates or glucocorticoids
* No pregnancy, breastfeeding, or planning to become pregnant during the study (diet group only)
* No lactose intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Change in the levels of cerebrospinal fluid (CSF) proopiomelanocortin (POMC) derived peptides (fmol/ml) that occur in subjects after diet induced weight loss compared to RYGB and SG. | Up to 12 months
  POMC plays a critical role in regulating energy balance and levels decrease in the hypothalamus after diet-induced weight loss; this may lead to weight regain after dieting.
Comparison of changes in the CSF proteome that occur after diet-induced weight-loss compared to RYGB and SG using unbiased proteomic analysis. | Up to 12 months

SECONDARY OUTCOMES:
Comparison of the changes in Agouti-related protein (AgRP) concentrations (fmol/ml) in CSF and plasma that occur in subjects after diet induced weight loss compared to RYGB and SG. | Up to 12 months
  AgRP is neuropeptide that stimulates food intake and increases after diet-induced weight loss.
Comparison of changes in CSF cortisol (ng/mL) that occur in subjects after diet induced weight loss compared to RYGB and SG. | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Wardlaw, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No